CLINICAL TRIAL: NCT02472405
Title: Comparing the 595/1064nm Multiplex Laser to the 595nm PDL in the Treatment of Surgical Scars in a Blinded, Randomized, Controlled Trial
Brief Title: Multiplex Laser vs. PDL (Pulsed Dye Laser ) in the Treatment of Surgical Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Keyvan Nouri, MD, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20140348
Record Dates: First submitted 2015-03-02; First posted 2015-06-15 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: Each participant scar was randomized to the 3 treatment arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 595nm PDL (Active Comparator): One third of the scar will be treated with 595nm PDL solely for 3 weeks (1 treatment session per week). A blinded observer will evaluate each third of the scar 4 weeks after the last treatment session using the POSAS system.
  Interventions: Device: 595nm PDL
- 595/1064nm Multiplex Laser (Active Comparator): One third of the scar will be treated with 595/1064nm Multiplex laser for 3 weeks (1 treatment session per week). A blinded observer will evaluate each third of the scar 4 weeks after the last treatment session using the POSAS system.
  Interventions: Device: 595/1064nm Multiplex Laser
- Control (No Intervention): One third of the scar will be left untreated for the duration of the study. A blinded observer will evaluate each third of the scar 4 weeks after the last treatment session using the POSAS system.

INTERVENTIONS:
Device: 595/1064nm Multiplex Laser — The multiplex cynergy laser will be used for this study. A third of the scar will solely be treated with the 595nm PDL.
  Arms: 595/1064nm Multiplex Laser
Device: 595nm PDL — One third of the scar will be treated with 595nm PDL solely for 3 weeks (1 treatment session per week).
  Arms: 595nm PDL

SUMMARY:
This study aims to determine if the 595nm Pulsed dye laser, the combined 595/1064nm Multiplex laser or no treatment results in a better outcome in the quality of the surgical scar using the multiplex cynergy laser, starting treatment the day of suture removal.

DETAILED DESCRIPTION:
This study aims to determine if the 595nm Pulsed dye laser, the combined 595/1064nm Multiplex laser or no treatment results in a better outcome in the quality of the surgical scar using the multiplex cynergy laser, starting treatment the day of suture removal.

Patients will be offered the opportunity of enrolling in the trial before their surgery. If they qualify and agree to participate they will sign informed consent and Health Insurance Portability and Accountability Act (HIPAA) form.

The surgical defect should be closed primarily, with the minimal scar length being 3cm. The scar will be randomized into 3 equal thirds, each third will randomly receive either: no treatment, 595nm PDL, or 595/1064nm Multiplex laser. A total of 3 laser treatments will be performed over a period of 3 weeks (one treatment session performed every week), and the patient will come in for a final follow up visit, for a final assessment of the scar using the Patient and Observer Scar Assessment Scale (POSAS) system.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin types 1-3
* Suture line should be at least 3 cm long

Exclusion Criteria:

* The patient should not be receiving any alternate systemic, topical or intralesional treatment of the scars during the study
* Pregnant or lactating females
* Fitzpatrick skin type 4-6
* A history of keloids or hypertrophic scars

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Nouri, MD, Principal Investigator — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 595nm PDL - 595/1064nm Multiplex - Control: A third of each participant's scar was treated with 595nm PDL solely for 3 weeks (1 treatment session per week). Another third of the scar was treated with 595/1064nm Multiplex laser for 3 weeks (1 treatment session per week). And the remaining third of the scar was left untreated for the duration of the study. The order of treatment was not randomized. A blinded observer evaluated each third of the scar 4 weeks after the last treatment session using the POSAS system.
Period: Overall Study
Arm/Group | 595nm PDL - 595/1064nm Multiplex - Control
Started | 18
Completed | 8
Not Completed | 10
Not completed — Lost to Follow-up | 9
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | 595nm PDL - 595/1064nm Multiplex - Control
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: POSAS (The Patient and Observer Scar Assessment Scale) Measure
Description: POSAS is a scale that contains the following parameters: pigmentation, vascularity, pliability, height, surface area, and patient input with regards to pain, itching, relief, stiffness, color and thickness. Both the patient and the observer are asked to give their Overall Opinion on the appearance of the scar. Again, a 10-point scale (ranging from 1 to 10) is used in which 10 corresponds to the worst imaginable scar.
Time Frame: 2 months
Population: The measurement used for this outcome was completed 4 weeks post final intervention, only eight participants completed the study protocol, but only 6 participant's POSAS score was collected. Observer's score for the POSAS is not available. Only the score for the participants was reported.
Measure: Mean (Standard Deviation); unit: Score
Groups:
- 595nm PDL: One third of the scar was treated with 595nm PDL solely for 3 weeks (1 treatment session per week). A blinded observer evaluated each third of the scar 4 weeks after the last treatment session using the POSAS system.
  595nm PDL: One third of the scar was treated with 595nm PDL solely for 3 weeks (1 treatment session per week).
- 595/1064nm Multiplex Laser: One third of the scar was treated with 595/1064nm Multiplex laser for 3 weeks (1 treatment session per week). A blinded observer evaluated each third of the scar 4 weeks after the last treatment session using the POSAS system.
  595/1064nm Multiplex Laser: The multiplex cynergy laser was used for this study. A third of the scar was solely be treated with the 595nm PDL.
- Control: One third of the scar was left untreated for the duration of the study. A blinded observer evaluated each third of the scar 4 weeks after the last treatment session using the POSAS system.
Arm/Group | 595nm PDL | 595/1064nm Multiplex Laser | Control
Number analyzed (Participants) | 6 | 6 | 6
Score | 2.5 (1.5) | 2.5 (1.5) | 2.5 (1.5)

ADVERSE EVENTS:
Time Frame: Seven weeks.
Groups:
- 595nm PDL - 595/1064nm Multiplex Laser - Control: A third of each participant's scar was treated with 595/1064nm Multiplex laser for 3 weeks (1 treatment session per week). Another third of the scar was treated with 595nm PDL solely for 3 weeks (1 treatment session per week). The remaining third of the scar was left untreated for the duration of the study. A blinded observer evaluated each third of the scar 4 weeks after the last treatment session using the POSAS system.
  595/1064nm Multiplex Laser: The multiplex cynergy laser will be used for this study. A third of the scar will solely be treated with the 595nm PDL.
Arm/Group | 595nm PDL - 595/1064nm Multiplex Laser - Control
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 595nm PDL - 595/1064nm Multiplex Laser - Control (N=18)
Minor bleeding and scabbing (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes